CLINICAL TRIAL: NCT00056875
Title: Safety and Efficacy of Recombinant Human Keratinocyte Growth Factor in Unrelated and Related Transplants
Brief Title: Recombinant Human Keratinocyte Growth Factor in Unrelated and Related Transplants
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Non-Randomized | Masking: None | Purpose: Prevention
Other Study IDs: 2146
Record Dates: First submitted 2003-03-25; First posted 2003-03-27 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2006-02

CONDITIONS: Graft Versus Host Disease
Keywords: graft versus host disease; bone marrow transplant; alternative donor
MeSH Terms: conditions — Graft vs Host Disease | interventions — Fibroblast Growth Factor 7

INTERVENTIONS:
Drug: recombinant human keratinocyte growth factor

SUMMARY:
This is a single arm dose escalation study of recombinant human keratinocyte growth factor given to patients undergoing allogeneic bone marrow transplantation who are at high risk for graft versus host disease (GVHD).

DETAILED DESCRIPTION:
Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
Eligible for full intensity bone marrow transplant (BMT) conditioning but who lack a 6/6 HLA idential sibling donor

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2002-09; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: John Levine, MD, Principal Investigator — Univeristy of Michigan
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States